CLINICAL TRIAL: NCT07278037
Title: A Retrospective Analysis of the Longitudinal Pattern of Tranexamic Acid Administration in Parturients Undergoing Cesarean Delivery Complicated by Postpartum Hemorrhage
Brief Title: Trends in the Administration of Tranexamic Acid for Postpartum Hemorrhage
Status: Recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 776/2568(IRB3); Si 717/2025 (Other: Faculty of Medicine Siriraj Hospital Mahidol University)
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Hemorrhage; Delivery Complication; Cesarean Section Complications; Perinatal Problems
Keywords: cesarean delivery; complications; postpartum hemorrhage; tranexamic acid
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tranexamic acid group: Patients received tranexamic acid after postpartum hemorrhage
  Interventions: Drug: Tranexamic acid
- Non tranexamic acid group: Patients did not receive tranexamic acid after postpartum hemorrhage

INTERVENTIONS:
Drug: Tranexamic acid — The number of patients received tranexamic acid after postpartum hemorrhage
  Other Names: TXA
  Groups: Tranexamic acid group

SUMMARY:
Postpartum hemorrhage (PPH) is the global leading cause of maternal death, with 20-30% of maternal deaths in Thailand linked to hemorrhage. The WOMAN Trial (2017) provided strong evidence that administering tranexamic acid (TXA)within three hours of bleeding onset lowered PPH-related mortality by 31%. Consequently, the World Health Organization (WHO) updated its guidelines, recommending TXA as part of the standard treatment package for all PPH cases. Following this, the use of TXA has been widely adopted globally and increased in Thailand. A recent study at a major Thai university hospital observed a significant increase in TXA administration after 2017. The current study aims to further analyze the recent growth rate of TXA use and its impact on obstetric and perinatal outcomes during cesarean deliveries with PPH.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is the foremost global cause of maternal mortality and represents a critical public health challenge. While the frequency of PPH varies worldwide, its prevalence remains markedly higher in developing nations. For instance, in Thailand, maternal death rates were reported between 20.0 and 40.5 per 100,000 deliveries from 1990 to 2015, with PPH accounting for 20% to 30% of these fatalities. Standard care for PPH involves fluid resuscitation, vital sign monitoring, uterotonic medications, and various non-surgical or surgical procedures. Within this framework, tranexamic acid (TXA), an antifibrinolytic agent, has gained substantial clinical recognition as an effective pharmacological treatment for PPH.

The therapeutic utility of TXA was strongly validated by the pivotal World Maternal Antifibrinolytic Trial (WOMAN Trial), a large international randomized controlled trial published in 2017. This landmark study definitively showed that administering TXA within three hours of bleeding onset resulted in a statistically significant 31% reduction in mortalityspecifically related to hemorrhage in PPH cases. This compelling evidence immediately prompted the World Health Organization (WHO) to update its clinical recommendations. The revised WHO guideline now advocates for the use of TXA as soon as possible in all PPH cases, regardless of the delivery method, integrating it into the standard comprehensive treatment protocol.

In the wake of this influential global recommendation, numerous healthcare systems and clinical institutions have revised their PPH management algorithms to incorporate TXA. Consequently, the utilization of tranexamic acid has demonstrably increased across several countries, including Thailand. A recent secondary analysis conducted at a major Thai university hospital, which reviewed 649 PPH cases following cesarean deliveries (2016-2020), confirmed a statistically significant surge in TXA administration after the 2017 WHO guideline change. Although patients receiving TXA were typically those with a greater history of antepartum hemorrhage and significantly higher measured blood loss, the study noted no corresponding change in adverse maternal outcomes, such as rates of blood transfusions, massive hemorrhage, hysterectomy, or intensive care unit admissions.

The present study aims to further analyze and update the data, specifically delineating the recent temporal trend in TXA administration and thoroughly evaluating the comprehensive influence of the WHO recommendations on local obstetric hemorrhage management and associated perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients underwent cesarean delivery with primary postpartum hemorrhage

Exclusion Criteria:

1. Gestational age at less than 24 weeks
2. Absence of the anesthetic record
3. Received tranexamic acid in the antepartum period
4. Blood loss less than 1,000 ml

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients underwent cesarean delivery with diagnosis of primary postpartum hemorrhage at Siriraj Hospital, Bangkok, Thailand
Sampling Method: Non-Probability Sample
Enrollment: 648 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of tranexamic acid administration divided by year | Within 24 hours after delivery
  Number of patients received tranexamic acid after diagnosis of postpartum hemorrhage

SECONDARY OUTCOMES:
Quantity of blood loss | Within 24 hours after delivery
  Quantity of blood loss recorded in patients chart
Number of patients received blood transfusion | Within 24 hours after delivery
  Number of patients received packed red cells transfusion
Number of patients received additional obstetrical interventions | Within 24 hours after delivery
  Number of patients received additional obstetrical interventions such as intrauterine balloon insertion, hysterectomy, uterine artery ligation, B-lynch suture
Number of patients receive reoperation | Within 24 hours after delivery
  Reoperation within 24 hours after cesarean delivery
Causes of postpartum hemorrhage | Within 24 hours after delivery
  Causes of postpartum hemorrhage divided into 4 categories, 1: uterine atony; 2: abnormal placentation; 3: trauma to internal organ(s); 4:abnormal coagulation
Factors influencing tranexamic acid administration | Within 24 hours after delivery
  Identify factors influencing tranexamic acid administration eg. history of antepartum hemorrhage, placental cause of PPH etc.
Side effect of tranexamic acid administration | After delivery to 30 days
  Side effect of tranexamic acid administration eg. thromboembolism, stroke
Hospital length of stay | After delivery to 30 days
  Hospital length of stay in days
Maternal Mortality | After delivery to 30 days
  Maternal death rate if death occur

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
The plan is undecided